CLINICAL TRIAL: NCT00844376
Title: An Open Label, Single Dose, Randomized 2-Way Crossover Study To Estimate The Relative Bioavailability Of Atorvastatin Commercial Tablet, And An Extemporaneous Preparation (EP) Suspension Formulation, In Healthy Subjects
Brief Title: Bioavailability Study for New Atorvastatin Formulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A2581164
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Results first posted 2009-10-21 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Hypercholesterolemia
Keywords: Cardiovascular Diseases
MeSH Terms: conditions — Hypercholesterolemia; Cardiovascular Diseases | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Other): Extemporaneous preparation suspension Atorvastatin prototype formulation
  Interventions: Drug: Atorvastatin suspension
- Reference (Other): Commercial atorvastatin tablet (Lipitor®)
  Interventions: Drug: Lipitor

INTERVENTIONS:
Drug: Atorvastatin suspension — A single dose of 80 mg Atorvastatin suspension
  Arms: Test
Drug: Lipitor — A single dose of 80 mg Lipitor tablet
  Other Names: Atorvastatin
  Arms: Reference

SUMMARY:
The purpose of this study is to estimate the relative bioavailability of the commercial tablet with one prototype extemporaneous preparation suspension formulation, to assist with internal decision making on formulation development.

DETAILED DESCRIPTION:
Estimation of Relative Bioavailability

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects
* Body Mass Index (BMI) of approximately 18 to 30 kg/m2

Exclusion Criteria:

* Any condition possibly affecting drug absorption
* A positive urine drug screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581164&StudyName=Bioavailability%20Study%20for%20New%20Atorvastatin%20Formulation

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One center in the U.S.
Pre-assignment Details: This study contained two sequences of 6 subjects per sequence. Each sequence received either test treatment followed by reference treatment, or reference treatment followed by test treatment. The order of administration was randomized to either of 2 sequences.
Groups:
- Test Drug First (Atorvastatin EP Suspension): 80-milligram (mg) Extemporaneous preparation (EP) suspension atorvastatin prototype formulation as a single dose in the first intervention period and commercial (reference) 80 mg atorvastatin tablet (Lipitor®) as a single dose in the second intervention period. Period 2 began immediately after period 1.
- Reference Drug First (Atorvastatin Tablet): 80-mg Commercial atorvastatin tablet (Lipitor®) as a single dose in the first intervention period and 80-mg EP suspension atorvastatin prototype formulation as a single dose in the second intervention period. Period 2 began immediately after period 1.
Period: Period 1: First Intervention
Arm/Group | Test Drug First (Atorvastatin EP Suspension) | Reference Drug First (Atorvastatin Tablet)
Started | 6 | 6
Completed | 5 | 6
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Period 2: Second Intervention
Arm/Group | Test Drug First (Atorvastatin EP Suspension) | Reference Drug First (Atorvastatin Tablet)
Started | 5 | 6
Completed | 5 (Total subjects administered Test drug = 12; total subjects administered Reference drug = 11.) | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Predose (Time Zero) to 48 Hours Post-dose (AUC48)
Description: Geometric means of AUC48 = area under the plasma concentration-time profile from time zero (0) to 48 hours postdose of atorvastatin (test versus [vs] reference); measured in nanograms times hour per milliliter (ng.hr/mL).
Time Frame: 5 days
Measure: Geometric Mean (Full Range); unit: ng.h/mL
Groups:
- Test: 80-mg Extemporaneous preparation suspension Atorvastatin prototype formulation
- Reference: 80-mg Commercial atorvastatin tablet (Lipitor®)
Arm/Group | Test | Reference
Number analyzed (Participants) | 12 | 11
ng.h/mL | 135.05 [52.5 to 233.00] | 140.79 [64.10 to 243.00]
Statistical Analysis 1: Comparison: Test vs Reference; Ratio of adjusted means (test/reference), and 90% CI for ratio--for AUC48; restricted (residual) maximum likelihood (REML) method of estimation; Test type: Superiority or Other; Mixed Models Analysis; The mixed effects model was implemented using SAS Proc Mixed, with REML estimation method and Kenward-Roger degrees of freedom algorithm; ratio of adjusted geometric means = 95.77, 90% CI [85.82 to 106.88] — Natural log transformed AUC48 was analyzed using a mixed effect model with sequence, period and treatment as a fixed effect and subject within sequence as a random effect

2. Primary Outcome: Area Under the Curve From Predose (Time Zero) to Extrapolated Infinite Time (AUC Infinity)
Description: Geometric means of AUC infinity (AUCinf) = area under the plasma concentration-time curve from time zero (0) extrapolated to infinite time; measured in ng.hr/mL of atorvastatin (test vs reference).
Time Frame: 5 days
Measure: Geometric Mean (Full Range); unit: ng.hr/mL
Arm/Group | Test | Reference
Number analyzed (Participants) | 12 | 11
ng.hr/mL | 135.88 [51.20 to 234.00] | 142.86 [65.00 to 247.00]
Statistical Analysis 1: Comparison: Test vs Reference; Ratio of adjusted means (test/reference), and 90% CI for ratio--for AUCinf; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; ratio of adjusted geometric means = 95.04, 90% CI [84.99 to 106.27] — Natural log transformed AUCinf was analyzed using a mixed effect model with sequence, period and treatment as a fixed effect and subject within sequence as a random effect

3. Secondary Outcome: Area Under the Curve From Predose (Time Zero) to Last Quantifiable Concentration (AUClast)
Description: Geometric mean of AUClast = area under the plasma concentration-time curve from time zero (0) to the last measurable concentration of atorvastatin (test vs reference); measured as ng.hr/mL
Time Frame: 5 days
Measure: Geometric Mean (Full Range); unit: ng.hr/mL
Arm/Group | Test | Reference
Number analyzed (Participants) | 12 | 11
ng.hr/mL | 130.21 [45.50 to 231.00] | 137.49 [56.00 to 243.00]
Statistical Analysis 1: Comparison: Test vs Reference; Ratio of adjusted means (test/reference), and 90% CI for ratio--for AUClast; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; ratio of adjusted geometric means = 94.86, 90% CI [83.86 to 107.29] — Natural log transformed AUClast was analyzed using a mixed effect model with sequence, period and treatment as a fixed effect and subject within sequence as a random effect

4. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Geometric mean of Cmax = maximum observed plasma concentration of atorvastatin (test vs reference); measured in nanograms per milliliter (ng/mL).
Time Frame: 5 days
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | Test | Reference
Number analyzed (Participants) | 12 | 11
ng/mL | 38.74 [20.30 to 86.80] | 33.24 [16.60 to 52.20]
Statistical Analysis 1: Comparison: Test vs Reference; Ratio of adjusted means (test/reference), and 90% CI for ratio--for Cmax; Test type: Superiority or Other; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; ratio of adjusted geometric means = 117.90, 90% CI [98.22 to 141.53] — Natural log transformed Cmax was analyzed using a mixed effect model with sequence, period and treatment as a fixed effect and subject within sequence as a random effect

5. Secondary Outcome: Terminal Phase Rate Constant (Kel)
Description: Geometric mean of Kel= termination phase rate constant for atorvastatin (test vs reference); measured as 1 per hour (1/hr).
Time Frame: 5 days
Measure: Geometric Mean (Full Range); unit: 1/hr
Arm/Group | Test | Reference
Number analyzed (Participants) | 12 | 11
1/hr | 0.12 [0.09 to 0.26] | 0.10 [0.06 to 0.15]

6. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax)
Description: Median of Tmax = time to maximum plasma concentration (Cmax) (test vs reference); measured in hours (hr).
Time Frame: 5 days
Measure: Median (Full Range); unit: hr
Arm/Group | Test | Reference
Number analyzed (Participants) | 12 | 11
hr | 0.52 [0.50 to 2.00] | 0.50 [0.50 to 3.00]

7. Secondary Outcome: Plasma Elimination Half-life (t1/2)
Description: Mean of t1/2 = terminal elimination half-life of atorvastatin (test vs reference); measured in hours.
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Test | Reference
Number analyzed (Participants) | 12 | 11
hr | 5.95 (1.40) | 7.21 (2.23)

ADVERSE EVENTS:
Arm/Group | Test | Reference
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 1/12 | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test (N=12) | Reference (N=11)
headache (Nervous system disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.